CLINICAL TRIAL: NCT07362485
Title: Indocyanine Green Guided Identification of Sentinel Lymph Nodes Via Mastectomy Incision in Breast Cancer Patients (INIGMA Study)
Brief Title: Finding Sentinel Lymph Nodes During Mastectomy Using Indocyanine Green (INIGMA Study)
Acronym: INIGMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Henskens (Other)
Collaborators: Isala (Other)
Responsible Party: Sponsor-Investigator, Isabelle Henskens, Coordinating investigator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL80591.100.22
Record Dates: First submitted 2026-01-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Sentinel Lymph Node Biopsy (SLNB); Sentinel Lymph Node Detection; Sentinel Lymph Node; Lymphatic Metastasis; Fluorescence Imaging; Indocyanine Green (ICG); Radioisotopes; Lymph Node Mapping; Mastectomy
Keywords: Breast cancer; Sentinel lymph node biopsy; Indocyanine green; Mastectomy; Fluorescence imaging; Lymph node mapping; Surgical oncology; Techetium nanocolloïd; Radioisotope
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: All participants receive both indocyanine green (ICG) fluorescence imaging and standard 99mTc-nanocolloid sentinel lymph node mapping during the same surgical procedure. The procedure is primarily performed using ICG fluorescence imaging, with 99mTc serving as the control method to assess the diagnostic performance of ICG compared to 99mTc. Each patient serves as her own control in this within-subject comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG-fluorescence imaging with 99mTc control for SLNB (Experimental): This experimental arm involves participants receiving indocyanine green (ICG) fluorescence imaging as the primary method for sentinel lymph node biopsy (SLNB), with 99mTc-nanocolloid serving as the within-patient control. Both methods are applied during the same surgical procedure. This design allows each participant to serve as their own control for comparing the diagnostic perfomance of both techniques directly in indentifying sentinel lymph nodes via mastectomy incision.
  Interventions: Other: Indocyanine green (ICG)-fluorescence guided sentinel lymph node biopsy

INTERVENTIONS:
Other: Indocyanine green (ICG)-fluorescence guided sentinel lymph node biopsy — ICG-fluorescence is used as the primary tracer to identify SLNs during SLNB in breast cancer surgery. The standard 99mTc-nanocolloid method is used as a control to verify the sentinel lymph nodes identified by ICG. Surgeons are blinded to preoperative lymphoscintigraphy results. After general anesthesia, 5 mg (2 mL of 2.5 mg/mL solutio) of ICG is injected sub-/intracutaneous periareolarly. ICG-fluorescence is detected using near-infrared imaging. SLNB via mastectomy incision is performed. The most fluorescent lymph node is excised first, followed by (maximal 2) additional fluorescent nodes. The excised nodes are tested for 99mTc-activity using a gamma probe. The axilla is then checked with the gamma probe and and palpation for any remaining nodes, which are excised if their radiation count exceeds 10% of the hottest node. All excised lymph nodes are sent for pathological examination to determine the presence of cancer cells. After surgery, the lymphoscintigraphy results are announced.

SUMMARY:
This pilot study evaluates the diagnostic value of indocyanine green (ICG) fluorescence for sentinel lymph node biopsy (SLNB) performed through the mastectomy incision in breast cancer patients.

Women with clinically node-negative, invasive T1-T3 breast cancer undergoing mastectomy with SLNB at St. Antonius or Isala Hospital will be included. All patients receive standard 99mTc injection preoperatively, followed by 5 mg (2mL) ICG injection after anesthesia. The axilla will be explored for fluorescent lymph nodes via the mastectomy incision, avoiding a separate axillary incision.

Primary outcome: ICG detection rate for SLN identification via the mastectomy incision.

Secondary outcomes: Comparison with 99mTc detection, number of nodes identified, concordance between methods, pathology differences, detection time, and complications.

ICG is safe, non-ionizing, and causes no extra discomfort or visits. Risks and burden are minimal.

DETAILED DESCRIPTION:
Background:

Identifying lymphatic metastases is an important prognostic factor in the survival rate of breast cancer and the presence of lymphatic metastases carries consequences for further treatment. Results the non-inferiority INFLUENCE study and previous literature, led to the implementation of ICG-guided SLNBs via axillary incision as standard of care at the St. Antonius Hospital. The diagnostic performance of ICG-fluorescence for SNLBs using the mastectomy incision has not been described yet. Surgeons may perform SLNBs using the same incision as the mastectomy, rather than using an additional axillary incision. In such setting, extended operating distance and visualization with an improper angle might introduce challenges to identify the SLN by tracking lymphatic vessels into the axilla.

Objective:

This pilot study aims to identify the diagnostic value of indocyanine green (ICG) fluorescence imaging for SLNBs via the mastectomy incision.

Study design:

This is a multicenter, cross-sectional pilot study identifying the diagnostic value of indocyanine green (ICG) fluorescence imaging for SLN mapping via the mastectomy incision (different surgical approach).

Study population:

Women with breast cancer who are admitted to the St. Antonius Hospital or Isala Hospital. Inclusion criteria include clinically nodenegative, invasive T1-T3 breast cancer conformed by biopsy, preoperative axillary ultrasound to confirm clinical node-negative status and indication for mastectomy with SLN procedure.

Intervention:

All included patients will receive standard of care implying 99mTc injection the day before surgery. Consequently, 5 mg (2 ml) ICG will be injected periareolar after administration of general anaesthesia and before incision. The lateral edge of the standard mastectomy incision will be used to explore the axilla for ICG fluorescent lymph nodes to avoid a separate axillary incision. Then the excised nodes are tested for 99mTc activity with the standard gamma detecting probe as control. Lastly, the axilla will be explored with the standard gamma-probe for residual lymph nodes, and by common sight and palpation as a control.

Outcomes:

Primary: to assess the detection rate of the ICG method to identify the SLN via a mastectomy incision.

Secondary:

* The detection rate of 99mTc
* The difference in detection rate between ICG and 99mTc
* The median number of SLN identified with ICG and the standard 99mTc
* Percentage of SLNs that is fluorescent, but not positive for 99mTc
* Percentage of SLNs that are not fluorescent but positive for 99mTc
* The difference in pathology of the SLN found by ICG and 99mTc, including the difference between micro- and macro metastases (Mic and Mac resp.) and isolated tumor cells (ITCs)
* Detection time for the use of ICG to detect the SLN, defined as time between skin incision and SLN resection in minutes
* Complications, including wound infection, bleeding and lymphedema, of the combination of the ICG method and the standard 99mTc method to identify the SLN in mastectomies
* The number of serious adverse events from the combination of ICG and 99mTc

Risks and burden:

Consenting patients will not need to do anything extra than the standard of care outside signing the informed consent. Administration of ICG will be done while under general anaesthesia, so patients will not experience extra discomfort, neither do they need extra site visits as the follow-up will be done during the standard follow-up appointment. ICG is safe to use: it is nonionizing and knows little to no complications and adverse events. Considering the cut-off of 2 additional nodes, the preferable topographic location of these nodes and the clinical experience with additional lymph node sampling, no increase in risk of surgical morbidity is expected. Patients might benefit from the intervention as ICG can increase the identification rate of the sentinel lymph node procedure and might even replace 99mTc for SLN mapping. Thus, both risks and burden are minimal.

ELIGIBILITY:
Inclusion Criteria:

* Clinically node-negative, DCIS, invasive T1- T3 breast cancer confirmed by biopsy.
* Preoperative axillary ultrasound to confirm clinical node-negative status.
* Indication (or preference) for mastectomy and simultaneous SLN procedure.
* Written informed consent according to ICH/GCP and national regulations.

Exclusion Criteria:

* Patients < 18 years old
* Breast conserving surgery
* Direct reconstruction (with autologous tissue or implant)
* Known allergy for indocyanine green (ICG) or radioisotope technetium (99mTc), intravenous contrast or iodine
* Other concurrent solid tumour
* Hyperthyroidism or thyroid cancer
* Pregnancy or breast feeding
* Psychological, familial, sociological or geographical factors that could potentially hamper compliance with the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Identification rate of sentinel lymph nodes using indocyanine green fluorescence | During the surgical procedure (from skin incision to completion of sentinel lymph node resection)
  The identification rate is defined as the proportion of participants in whom at least one sentinel lymph node (SLN) is successfully identified using indocyanine green (ICG) fluorescence imaging via the mastectomy incision during surgery.

SECONDARY OUTCOMES:
Identification rate of sentinel lymph nodes using 99mTc | During the surgical procedure (from skin incision to completion of sentinel lymph node resection)
  The identification rate is defined as the proportion of participants in whom at least one sentinel lymph node is identified using the standard-of-care radioisotope technetium-99m (99mTc) during the same surgical procedure.
Difference in sentinel lymph node detection rate between ICG and 99mTc | During the surgical procedure (from skin incision to completion of sentinel lymph node resection)
  The absolute difference in identification rates between indocyanine green (ICG) fluorescence imaging and technetium-99m (99mTc) for sentinel lymph node detection within the same participant.
Number of sentinel lymph nodes identified per participant by ICG and 99mTc | During the surgical procedure (from skin incision to completion of sentinel lymph node resection)
  The total number of sentinel lymph nodes identified per participant using indocyanine green (ICG) fluorescence imaging and using technetium-99m (99mTc) during surgery.
Proportion of participants with fluorescent sentinel lymph nodes among those identified by 99mTc | During the surgical procedure (from skin incision to completion of sentinel lymph node resection)
  The percentage of participants in whom sentinel lymph nodes identified by the standard-of-care technetium-99m (99mTc) are also fluorescent when assessed with indocyanine green (ICG).
Fluorescent sentinel lymph nodes not positive for 99mTc | During the surgical procedure (from skin incision to completion of sentinel lymph node resection)
  The percentage of sentinel lymph nodes that demonstrate fluorescence with indocyanine green (ICG) but show no detectable activity on technetium-99m (99mTc) assessment.
Sentinel lymph nodes positive for 99mTc but not fluorescent | During the surgical procedure (from skin incision to completion of sentinel lymph node resection)
  The percentage of sentinel lymph nodes that are positive for technetium-99m (99mTc) activity but do not demonstrate fluorescence with indocyanine green (ICG).
Pathological status of sentinel lymph nodes identified by ICG and 99mTc | From surgical resection of sentinel lymph nodes until completion of histopathological assessment, assessed within approximately 3 weeks after surgery
  Pathological assessment of sentinel lymph nodes identified by indocyanine green (ICG) and technetium-99m (99mTc), including the presence of isolated tumour cells, micrometastases, or macrometastases.
Detection time for sentinel lymph node identification using ICG | During the surgical procedure (from skin incision to sentinel lymph node resection)
  Detection time is defined as the time in minutes between skin incision and resection of the first sentinel lymph node identified using indocyanine green (ICG) fluorescence imaging.
Procedure-related complications associated with ICG and 99mTc | From surgery up to 2 months postoperatively
  The proportion of participants experiencing complications related to the sentinel lymph node procedure using indocyanine green (ICG) and technetium-99m (99mTc), including seroma requiring drainage, wound infection requiring antibiotic or surgical treatment, bleeding requiring reoperation, and mild allergic reactions.
Serious adverse events related to ICG and 99mTc | From surgery up to 2 months postoperatively
  The number of participants experiencing serious adverse events related to indocyanine green (ICG) or technetium-99m (99mTc), including severe allergic reactions, death, or other serious adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Isala, Zwolle, Overijssel
  - St. Antonius Ziekenhuis, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
At present, there is no final decision regarding sharing of individual participant data (IPD). Data sharing will depend on ethical approval, participant consent, and compliance with applicable privacy regulations. If IPD sharing is pursued, only de-identified datasets relevant to the research question will be made available upon reasonable request to qualified researchers, under a data use agreement ensuring confidentiality and scientific integrity